CLINICAL TRIAL: NCT06478784
Title: Effects of Resistance Training in Multiple Sclerosis: a Randomized Trial. ACTIVE (Physical Activity and Its Impact on Patients With Multiple Sclerosis.)
Brief Title: Effects of Resistance Training in Multiple Sclerosis: a Randomized Trial.
Acronym: ACTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Collaborators: European University Miguel de Cervantes (Other)
Responsible Party: Principal Investigator, Alba Chavarria, Alba Chavarria Miranda, MD, Hospital Clínico Universitario de Valladolid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI-GR-23-3292
Record Dates: First submitted 2024-05-01; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis
Keywords: physical exercise; resistance training; neurofilaments; GFAP
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: We will include patients with multiple sclerosis in the ACTIVE GROUP (resistance training) and patients with multiple sclerosis CONTROL GROUP (low intensity aerobic training).
Who Masked: Participant, Investigator
Masking Description: A double-blind system will be maintained in which the exploring neurologists and the patient will not know the assigned therapeutic group. Randomly assigned to one or the other group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTIVE GROUP: Resistance training (Experimental): The experimental group (ACTIVE GROUP) will perform a circuit-based muscular strength program at high intensity, three days per week for 10 weeks.
  Interventions: Other: Resistance training
- CONTROL GROUP: Low intensity aerobic training (Active Comparator): Patients assigned to this CONTROL GROUP will perform exercise in static bicycle.They will perform aerobic training at low-moderate intensity (50% of the maximum power developed in cycloergometer) for 45 minutes three days a week, with a duration of 10 weeks.
  Interventions: Other: Low aerobic training

INTERVENTIONS:
Other: Resistance training — The experimental group (ACTIVE GROUP) will perform a circuit-based muscular strength program at high intensity three days per week for 10 weeks.
  Each session will last approximately 45 minutes.
  The Resistance training program will be supervised by staff from the Department of Health Sciences and Sports of the Miguel de Cervantes European University of Valladolid and will be carried out at the facilities of the Miguel de Cervantes European University of Valladolid.
  Arms: ACTIVE GROUP: Resistance training
Other: Low aerobic training — Patients assigned to this group will perform exercise in static bicycle during 45 minutes three days a week, with a duration of 10 weeks.
  This second group, despite performing the aerobic exercise, is considered control, since they will perform low-intensity aerobic exercise (50% of the maximum power developed in cycloergometer)
  The Resistance training program will be supervised by staff from the Department of Health Sciences and Sports of the Miguel de Cervantes European University of Valladolid and will be carried out at the facilities of the Miguel de Cervantes European University of Valladolid.
  Arms: CONTROL GROUP: Low intensity aerobic training

SUMMARY:
This is a longitudinal study to examine the effects of a short-term training program on neurofilamet and GFAP plasma levels. Participants will be divided in two groups: control group (moderate aerobic training) and active group (resistance training). The change in biomarkers will be analyzed pre and post intervention in both groups. Differences between groups will be also evaluated by investigators.

DETAILED DESCRIPTION:
Multiple sclerosis is a dysimmune and neurodegenerative disease of the central nervous system. Despite highly effective drug, multiple sclerosis represents the main cause of non-traumatic disability in young people. Interventions based on physical exercise have a positive impact on the course of the disease, although the pathophysiological mechanisms responsible for this benefit remain unknown. This project aims to investigate the impact of physical exercise on neuronal destruction in patients with multiple sclerosis.

To do this, the investigators will study the evolution of the concentrations of two markers of neuronal injury, acidic gliofibrillary protein (GFAP) and light chain neurofilaments (Nfl) in two groups of patients: a control group and a second group subjected to a supervised resistance physical exercise program performed during 10 weeks. Marker values will be compared before and after the intervention and between groups. The results will allow the investigators to delve into the pathophysiology of multiple sclerosis and the mechanism through which physical exercise impacts on the disease. In addition, the investigators will generate knowledge that will allow us to reinforce the idea of integrating physical exercise as part of the treatment in multiple sclerosis.

Project within the framework of the GRS(Gerencia Regional de Salud, Castilla y Léon) 28/10/A1/2023

ELIGIBILITY:
Inclusion Criteria:

1. - Diagnosis of multiple sclerosis according to the 2017 Mc Donald criteria (Thompson A et al).
2. - Age > 18 years - up to no age limit
3. - Disability assessed by the EDSS (Expanded disability status scale) with a score less than or equal to 4.
4. - Clinical stability. Not having had an outbreak of the disease in the last 6 months.
5. - No changes in the disease-modifying treatment in the last 6 months or no treatment.
6. - Radiological stability. Patients with last MRI (magnetic resonance imaging) performed without inflammatory activity (absence of new lesions on T2 sequences or lesions that enhance with gadolinium).
7. - They must sign the informed consent

Exclusion Criteria:

1. - Patients with a high level of physical activity according to the International Physical Activity Questionnaire(IPAQ) or latest WHO (World Health Organization) recommendations on physical activity
2. - Pregnant or breastfeeding patients.
3. - Concomitant pathologies that limit the performance of physical exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of plasma light chain neurofilaments (Nfl) level | 10 Weeks
  To evaluate the change of plasma neurofilament concentrations (pg/mL) between the two groups of multiple sclerosis patients, the control group that will perform moderate aerobic exercise vs. the group subjected to the resistance training intervention.

SECONDARY OUTCOMES:
Comparison of plasma Glial fibrillary acidic protein (GFAP) level | 10 weeks
  To study the change of plasma Glial fibrillary acidic protein (GFAP)(pg/mL) between the two groups of multiple sclerosis patients, the control group that will perform moderate aerobic exercise vs. the group subjected to the resistance training intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alba Chavarria Miranda, MD, Principal Investigator — Hospital Clínico Universitario de Valladolid
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mulero P, Maroto-Izquierdo S, Redondo N, Gonzalo-Benito H, Chavarria-Miranda A, Calvo H, Cabero MI, Hernandez M, Nieto ML, Tellez N. Effect of resistance exercise training on plasma neurofilaments in multiple sclerosis: a proof of concept for future designs. Neurol Sci. 2023 Nov;44(11):3997-4000. doi: 10.1007/s10072-023-06896-5. Epub 2023 Jun 19. PMID 37335403